CLINICAL TRIAL: NCT04916587
Title: Supporting the Implementation of a State Policy on Screening for Adverse Childhood Experiences (ACEs) in Federally Qualified Health Centers (FQHC)
Brief Title: Implementation of Adverse Childhood Experiences (ACEs) Policy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 22-0547; R21MH123835 (NIH)
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Adverse Childhood Experiences
Keywords: Well-child screening; Implementation science

STUDY DESIGN:
Intervention Model Description: [Update May/2024] We conduct a stepped wedge, cluster pragmatic trial without transition periods. Three clinics (clusters) receive the intervention at different points in time. The full trial lasts 18 months, conducted in seven extended 10-week periods. Control status refers to clinics following standard care. During the COVID-19 pandemic, clinics did not start ACEs screenings. Intervention status refers to clinics experiencing the implementation strategy and ACEs screenings. During baseline (weeks 1-10), we collect pre-implementation data on mental health referrals, and child socio-demographics. Following baseline, clinics receive the intervention in six steps. Outcomes collected in week 10/each step
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACEs Screenings and a Multifaceted Implementation Strategy (Active Comparator): [Update May/2024] ACEs pediatric screenings in primary care settings. This study will focus on screening children ages 0-5, in line with the partnering FQHC's ACEs screening priorities. The implementation strategy components are: 1) video-trainings for clinic personnel (care team staff and providers); 2) technical implementation support to increase inner context capacity, 3) use of a validated clinical screening tool - Pediatric Symptoms Checklist (PSC-17), used in pediatric settings to assess behavioral and social/emotional development. For this study, we use the PSC tools that are tailored to children ages 0 to 5 years old with the Baby Pediatric Symptomatology Checklist (BPSC) for ages 0 to 18 months, and the Preschool Pediatric Symptom Checklist (PPSC) for ages 18 to 60 months. This screening tool is needed as the PEARLS only assesses ACEs exposure; and 4) use of a technology-based tailored ACEs algorithm that incorporates multiple data sources.
  Interventions: Other: Implementation Strategy of ACEs Screenings
- Standard Care (Other): Clinics provide standard care that includes unstructured conversations between clinicians and caregivers about the child(ren)'s needs and a service referral as needed.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Implementation Strategy of ACEs Screenings — We will use implementation mapping, guided by the EPIS framework, to promote a co-created process and refine the strategy comprised of online training videos, a customized ACEs algorithm and use of technology to improve workflow efficiency, implementation technical assistance/coaching, and written implementation protocols.
  Arms: ACEs Screenings and a Multifaceted Implementation Strategy
Other: Usual Care — The ACEs Aware policy goal is to "equip providers with training and clinical protocols to screen children and adults for ACEs, detect ACEs early, and connect patients to interventions, resources, and other support to improve patient health and well-being." ACEs screenings are comprised of: a) a 2-hour on-line provider training; b) the Pediatric ACEs and Related Life-events Screener or PEARLS tool; c) an ACEs associated health conditions checklist; and d) complete a wellness exam. The primary care provider uses multiple sources of information to identify a child's need for follow-up services.
  Other Names: ACEs Screenings
  Arms: Standard Care

SUMMARY:
Adverse Childhood Experiences (ACEs) are pervasive among children with 45% experiencing at least one ACE and 10% experiencing three or more, placing them at high risk for toxic stress and symptomatology. Yet, ACEs often go undetected in primary care settings during well-child visits due to unclear policies and tested implementation strategies. This pilot study will use mapping methodology, guided by the Exploration, Preparation, Implementation and Sustainment (EPIS) framework, to refine a multi-faceted strategy supporting the implementation of the state of California's 2020 policy promoting universal ACE screening in community clinics, and a stepped-wedge trial to test the impact of the strategy on implementation and child-level outcomes.

DETAILED DESCRIPTION:
Adverse Childhood Experiences (ACEs) are defined as traumatic events occurring before age 18, such as maltreatment, life-threatening accident, harsh migration experiences or exposure to violence. ACEs are pervasive, with 45% experiencing at least one ACE and 10% experiencing three or more ACEs, placing them at high risk for negative life outcomes. ACEs are more prevalent among minority and immigrant communities due to exposure to poverty, discrimination, community violence, national disasters, and refugee experiences. ACEs screenings have potential value in identifying children experiencing toxic stress and the physical and mental health conditions associated with it such as asthma, Attention Deficit Hyperactive Disorder (ADHD) and anxiety. Yet, they are seldom used in primary care during well-child visits. The Surgeon General of the state of California have addressed this care gap by issuing an ACEs screening policy. Starting January 2020, MediCal, California's Medicaid health care program, will reimburse primary care settings ($29) for using the Pediatric ACEs and Related Life-events Screener (PEARLS) tool to screen children for ACEs during wellness visits. Despite significant investment in California and nationwide, evidence of the public health value of universal child screening policies is unclear. Increased screening efforts often do not translate into higher access to care for children and may even exacerbate disparities by increasing stigma and reinforcing a deficit view of marginalized groups. These results have been attributed to a lack of rigorous studies testing implementation strategies suited for pediatric screening policies. This mixed-method study will fill this gap by refining and testing an implementation strategy using a multi-site controlled trial within a Federally Qualified Health Center in Southern California. [Update 05/2024] Using the EPIS framework, we will employ a hybrid (type 2), controlled trial using a stepped-wedge design (n=5 clinics; 3 in the study and 2 clinics already implementing ACEs and used as comparison sites) to test the central hypothesis that clinics employing a multifaceted implementation strategy will have higher fidelity and reach of the ACEs screening policy. The partner FQHC system experienced financial strain during the COVID-19 pandemic and several of the randomly selected clinics closed prior to randomization.Selection of replacement clinics was based on clinic capacity to participate in the trial. Secondary hypothesis: impact of the ACEs policy on child mental health service and symptom outcomes. Aims are: 1. Refine a multifaceted implementation strategy to support the implementation of the ACEs screening policy in community-based clinics, and 2. Pilot test the feasibility, acceptability, fidelity and reach of the implementation strategy and the impact of the ACEs policy on child patient-level outcomes. This project capitalizes on a rare opportunity to pilot test an implementation strategy to maximize the impact of a state-wide policy intended to improve child health in under-resourced settings.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 0-5 scheduled for wellness visit for upcoming week
* Caregiver of child is 18 years or older with legal custody or authority to arrange care for child
* Caregiver provides informed consent; signs consent form and HIPAA release form as well as coronavirus disease (COVID-19) information sheet
* Caregiver agrees to complete the Pediatric Symptoms Checklist or PSC
* Caregiver provides permission for socio-demographic information about their child to be pulled from EMR records, de-identified, and shared with PI

Exclusion Criteria:

* Children ages 0-5 scheduled for wellness visit for upcoming week
* Caregiver declines to provide signed informed consent, HIPAA release, or permission for socio-demographic data to be pulled from the Electronic Medical Records (EMR), de-identified and shared with PI; or declines to respond to 17 questions for the PSC
* Children ages 6-18 scheduled for wellness visits
* Children ages 0-5 scheduled for wellness visits outside the study data collection windows or at clinics not providing pediatric care
* Caregiver does not have legal guardianship or written authority to arrange care for the child

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7645 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Perez Jolles, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Borrego Health, Desert Hot Springs, California, United States

REFERENCES:
- [Derived] Jolles MP, Mack WJ, Rubio S, Helmkamp LJ, Saldana L, Aarons GA, Lau AS. Testing a multi-faceted strategy to support the implementation of ACEs screenings in primary care: results of a stepped-wedge pilot trial. Implement Sci Commun. 2025 Sep 1;6(1):92. doi: 10.1186/s43058-025-00771-4. PMID 40887671
- [Derived] Perez Jolles M, Mack WJ, Reaves C, Saldana L, Stadnick NA, Fernandez ME, Aarons GA. Using a participatory method to test a strategy supporting the implementation of a state policy on screening children for adverse childhood experiences (ACEs) in a Federally Qualified Health Center system: a stepped-wedge cluster randomized trial. Implement Sci Commun. 2021 Dec 20;2(1):143. doi: 10.1186/s43058-021-00244-4. PMID 34930500

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinics
Groups:
- Practice 1: This clinic was part of the study trial based on the seven extended 10-week periods in the Stepped Wedge schedule.
  Clinic 1: Baseline/Control for 10 weeks, followed by six intervention periods of 60 weeks total.
- Practice 2: This clinic was part of the study trial based on the seven extended 10-week periods in the Stepped Wedge schedule.
  Clinic 2: Baseline/Control for 20 weeks, followed by intervention period of 50 weeks total.
- Practice 3: This clinic was part of the study trial based on the seven extended 10-week periods in the Stepped Wedge schedule.
  Clinic 3: Baseline/Control for 30 weeks, followed by intervention period of 40 weeks total.
- Practice 4: This practice is a comparison group that did not receive the intervention throughout the study period.
- Practice 5: This is a comparison group that did not received the intervention
Period: Step 1: Months 1-2.3
Arm/Group | Practice 1 | Practice 2 | Practice 3 | Practice 4 | Practice 5
Started | 248; 1 Clinics | 587; 1 Clinics | 56; 1 Clinics | 351; 1 Clinics | 97; 1 Clinics
Completed | 248; 1 Clinics | 587; 1 Clinics | 56; 1 Clinics | 351; 1 Clinics | 97; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 2: Months 2.3 - 4.6
Arm/Group | Practice 1 | Practice 2 | Practice 3 | Practice 4 | Practice 5
Started | 367; 1 Clinics | 604; 1 Clinics | 74; 1 Clinics | 416; 1 Clinics | 151; 1 Clinics
Completed | 367; 1 Clinics | 604; 1 Clinics | 74; 1 Clinics | 416; 1 Clinics | 151; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 3: Months 4.6 - 6.9
Arm/Group | Practice 1 | Practice 2 | Practice 3 | Practice 4 | Practice 5
Started | 312; 1 Clinics | 470; 1 Clinics | 88; 1 Clinics | 322; 1 Clinics | 13; 1 Clinics
Completed | 312; 1 Clinics | 470; 1 Clinics | 88; 1 Clinics | 322; 1 Clinics | 13; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 4: Months 6.9 - 9.2
Arm/Group | Practice 1 | Practice 2 | Practice 3 | Practice 4 | Practice 5
Started | 189; 1 Clinics | 354; 1 Clinics | 75; 1 Clinics | 89; 1 Clinics | 0; 0 Clinics
Completed | 189; 1 Clinics | 354; 1 Clinics | 75; 1 Clinics | 89; 1 Clinics | 0; 0 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 5: Months 9.2 - 11.5
Arm/Group | Practice 1 | Practice 2 | Practice 3 | Practice 4 | Practice 5
Started | 238; 1 Clinics | 448; 1 Clinics | 100; 1 Clinics | 209; 1 Clinics | 0; 0 Clinics
Completed | 238; 1 Clinics | 448; 1 Clinics | 100; 1 Clinics | 209; 1 Clinics | 0; 0 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 6: Months 11.5 - 13.8
Arm/Group | Practice 1 | Practice 2 | Practice 3 | Practice 4 | Practice 5
Started | 260; 1 Clinics | 465; 1 Clinics | 97; 1 Clinics | 104; 1 Clinics | 0; 0 Clinics
Completed | 260; 1 Clinics | 465; 1 Clinics | 97; 1 Clinics | 104; 1 Clinics | 0; 0 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 7: Months 13.8 - 16.1
Arm/Group | Practice 1 | Practice 2 | Practice 3 | Practice 4 | Practice 5
Started | 227; 1 Clinics | 470; 1 Clinics | 106; 1 Clinics | 58; 1 Clinics | 0; 0 Clinics
Completed | 227; 1 Clinics | 470; 1 Clinics | 106; 1 Clinics | 58; 1 Clinics | 0; 0 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- Control: Clinics without implementing the strategy supporting ACEs screening.
- Interventions: Clinics started the ACEs screening and the implementation strategy.
- Comparison Clinics: Clinic starting ACEs screening without the implementation strategy
- Total: Total of all reporting groups
Arm/Group | Control | Interventions | Comparison Clinics | Total
Number analyzed (Participants) | 1657 | 4178 | 1810 | 7645
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1657 | 4178 | 1810 | 7645
  Between 18 and 65 years | NA — This study focused on screening children ages 0-5, in line with the partnering FQHC's ACEs screening priorities. | NA — This study focused on screening children ages 0-5, in line with the partnering FQHC's ACEs screening priorities. | NA — This study focused on screening children ages 0-5, in line with the partnering FQHC's ACEs screening priorities. | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — This study focused on screening children ages 0-5, in line with the partnering FQHC's ACEs screening priorities. | NA — This study focused on screening children ages 0-5, in line with the partnering FQHC's ACEs screening priorities. | NA — This study focused on screening children ages 0-5, in line with the partnering FQHC's ACEs screening priorities. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 788 | 2018 | 901 | 3707
  Male | 869 | 2160 | 909 | 3938
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 219 | 114 | 396
  Not Hispanic or Latino | 774 | 1719 | 718 | 3211
  Unknown or Not Reported | 820 | 2240 | 978 | 4038
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 774 | 1719 | 718 | 3211
  Black or African American | 63 | 219 | 114 | 396
  Other / Unknown | 820 | 2240 | 978 | 4038
Region of Enrollment [Number; unit: participants]
  United States | 1657 | 4178 | 1810 | 7645

OUTCOME MEASURES:

1. Primary Outcome: ACEs Screenings Reach
Description: The number of participants with ACEs screenings.
Time Frame: Every 10 weeks during the study trial, up to 19 months
Population: Children ages 0 - 5 years old attending the annual check-up visit at the clinic
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Interventions | Comparison Clinics
Number analyzed (Participants) | 1657 | 4178 | 1810
Participants | 0 | 468 | 73
Statistical Analysis 1: Comparison: Control; Test type: Superiority; Risk Difference (RD) = 11.6, 95% CI 2-sided [10.6 to 12.6]

2. Primary Outcome: Mental Health Service Referral
Description: Number of participants with a mental health referral (behavioral analysis, behavioral health, care coordinator, care management, child development/development center or social work)
Time Frame: Every 10 weeks during the study trial, up to 19 months.
Population: Children ages 0 - 5 years old attending the annual check-up visit at the clinic
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Interventions | Comparison Clinics
Number analyzed (Participants) | 1657 | 4158 | 1810
Participants | 6 | 302 | 4
Statistical Analysis 1: Comparison: Control; Test type: Superiority; Risk Difference (RD) = 7.5, 95% CI 2-sided [6.6 to 8.3]

3. Secondary Outcome: Changes in Baby Pediatric Symptoms (BPSS) / Preschool PSC (PPSC)
Description: The percentage of children screening positive for BPSS or PPSC from the time of the ACEs screening. These data were collected on a subsample of study participants during ACEs screenings (n=414). From that group, a total of 50 caregivers provided follow up information on PSC scores (n=50).
  This secondary outcome was collected as part of the strategy in the intervention group only (i.e., ACEs screenings plus the multifaceted implementation strategy group). The data were only collected from the "ACEs Screenings and a Multifaceted Implementation Strategy" Arm/Group.
Time Frame: First score measure during ACEs screenings. Follow-up scores from 8 - 16 months
Population: The PSC data was collected for a subset of the total sample. A group of caregivers reported on PSC scores during ACEs screenings (n=414). From that group, a total of 50 caregivers were randomly selected for follow-up to assess PSC scores after the screenings (n=50)
Measure: Count of Participants; unit: Participants
Groups:
- Follow up: PSC scores were collected after the ACEs screenings to assess differences between the intervention and follow up
Arm/Group | ACEs Screenings and a Multifaceted Implementation Strategy | Follow up
Number analyzed (Participants) | 414 | 50
Participants | 111 | 6
Statistical Analysis 1: Comparison: ACEs Screenings and a Multifaceted Implementation Strategy; Test type: Superiority; p = 0.03, Mixed Models Analysis; Odds Ratio (OR) = 0.36, 90% CI 2-sided [0.14 to 0.89]

4. Secondary Outcome: Acceptability of the Strategy
Description: Self-reported 4-item instrument to evaluate acceptability of ACEs policy and implementation efforts. 5-pt Likert scale; average score of 4+ shows acceptability. Good internal consistency (α=0.83). Test-retest reliability r=0.83. At the end of the stepped-wedge schedule, clinical personnel were invited to participate in a survey to evaluate the acceptability of the strategy. These data were collected on a subsample of clinic personnel involved in the implementation of the ACEs screenings at the study clinical sites.
  This self-reported 4-item instrument to evaluate acceptability used a 5-point Likert scale for each item, ranging from 1 (Completely Disagree) to 5 (Completely Agree). The total score is calculated by summing the responses across all four items, which range from 4 to 20, with higher scores indicating greater acceptability.
Time Frame: End of data collection -End of period 7 in the stepped-wedge schedule
Population: Children ages 0 - 5 years old attending the annual check-up visit at the clinic
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Interventions | Comparison Clinics
Number analyzed (Participants) | 0 | 10 | 0
units on a scale |  | 2.98 (0.90) |

5. Secondary Outcome: Feasibility of the Strategy
Description: Self-reported 4-item instrument to evaluate the feasibility of implementation efforts. 5-pt Likert scale; average score of 4+ shows ACEs policy and implementation strategy perceived as feasible. Good internal consistency (α=0.89). Test-retest reliability r=0.88. At the end of the stepped-wedge schedule, clinical personnel were invited to participate in a survey to evaluate the feasibility of the strategy. These data were collected on a subsample of clinic personnel involved in the implementation of the ACEs screenings at the study clinical sites.
  This self-reported 4-item instrument to evaluate feasibility used a 5-point Likert scale for each item, ranging from 1 (Completely Disagree) to 5 (Completely Agree). The total score is calculated by summing the responses across all four items, which range from 4 to 20, with higher scores indicating greater feasibility.
Time Frame: End of data collection- End of Period 7 based on the Stepped-Wedge Schedule
Population: Children ages 0 - 5 years old attending the annual check-up visit at the clinic
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Interventions | Comparison Clinics
Number analyzed (Participants) | 0 | 10 | 0
units on a scale |  | 2.97 (0.92) |

ADVERSE EVENTS:
Time Frame: No adverse event data were collected during the 19-month study period.
Description: This is a minimum risk intervention and mortality risk is not applicable to this study. The meaning of the 'zeroes' reported refers to - All-Cause Mortality, Serious and Other Adverse Events were not monitored/assessed.
Groups:
- Intervention Group: ACEs Screenings and a Multifaceted Implementation Strategy: [Update May/2024] Clinical Intervention: ACEs pediatric screenings in primary care settings. This study will focus on screening children ages 0-5, in line with the partnering FQHC's ACEs screening priorities.
  Implementation Intervention: We will use implementation mapping, guided by the EPIS framework, to promote a co-created process and refine the strategy comprised of online training videos, a customized ACEs algorithm and use of technology to improve workflow efficiency, implementation technical assistance/coaching, and written implementation protocols.The implementation strategy components are: 1) video-trainings for clinic personnel (care team staff and providers); 2) technical implementation support to increase inner context capacity, 3) use of a validated clinical screening tool - Pediatric Symptoms Checklist (PSC-17), used in pediatric settings to assess behavioral and social/emotional development. For this study, we use the PSC tools that are tailored to children ages 0 to 5 years old with the Baby Pediatric Symptomatology Checklist (BPSC) for ages 0 to 18 months, and the Preschool Pediatric Symptom Checklist (PPSC) for ages 18 to 60 months. This screening tool is needed as the PEARLS only assesses ACEs exposure; and 4) use of a technology-based tailored ACEs algorithm that incorporates multiple data sources.
- Control Group: Standard Care: Clinics provide standard care that includes unstructured conversations between clinicians and caregivers about the child(ren)'s needs and a service referral as needed.
- Comparison Group: Two clinics implementing ACEs screenings on their own (i.e., they were not part of the study), without the study's implementation strategy.
Arm/Group | Intervention Group: ACEs Screenings and a Multifaceted Implementation Strategy | Control Group: Standard Care | Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-07-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT04916587/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT04916587/SAP_001.pdf
  • Informed Consent Form (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04916587/ICF_002.pdf